CLINICAL TRIAL: NCT05873673
Title: The Effect of Coenzyme Q10 on Bone Regeneration in Jaw Defect After Cyst Enculation: A Randomized Controlled Clinical Trial
Brief Title: Coenzyme Q10 and Dentoalveolar Cyst
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer of oral and maxillofacial surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cyst, Jaw
MeSH Terms: conditions — Jaw Cysts | interventions — coenzyme Q10; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coenzyme group (Active Comparator)
  Interventions: Drug: Coenzyme Q10
- control group (Placebo Comparator)
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Coenzyme Q10 — cystic jaw defect filled with coenzyme Q10 gel
  Arms: coenzyme group
Drug: control group — cystic jaw defect filled with placebo gel
  Arms: control group

SUMMARY:
10 patients in each group will undergo cyst removal under local anesthesia. After cyst removal, the cystic cavity will be filled with placebo gel in the control group or coenzyme gel in the coenzyme group.

Bone density and volume will be assessed by cone beam CT immediately postoperative and 6months later for all patients

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with critical-size jaw cysts
* Medically stable
* No cystic lesion recurrence

Exclusion Criteria:

* Cystic lesion recurrence
* Medical problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-11 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
bone density | 6 months
  measure the bone density of new bone in the cystic cavity at 6 months by cone beam CT

SECONDARY OUTCOMES:
bone volume | 6months
  measure the bone volume in the defect by cone beam CT at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt